CLINICAL TRIAL: NCT07159178
Title: Investigation of the Effect of Shoulder Problems on Balance in Patients With Hemiplegia After Stroke
Brief Title: The Effect of Shoulder Problems on Balance in Hemiplegic Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, EDA SALGUT, principal ınvestigator, Istanbul Aydın University
Other Study IDs: IstanbuIAU
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Hemiplegia; Stroke
Keywords: Hemiplegia; Stroke; Shoulder Pain; Balance; postural control
MeSH Terms: conditions — Hemiplegia; Stroke; Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemiplegic Patients With and Without Shoulder Pain: This group includes hemiplegic patients after stroke. Participants were divided into two subgroups according to the presence or absence of shoulder pain. Assessments included pain, balance, and shoulder joint range of motion.

SUMMARY:
Shoulder problems are among the most common complications in hemiplegic patients and may impair shoulder biomechanics, negatively affecting mobility, transfers, and self-care. This study aims to investigate whether shoulder problems influence balance in hemiplegic patients after stroke. Patients with a first-ever stroke diagnosis, sufficient cognitive function (Mini Mental State Examination score ≥24), no visual impairments, and aged between 40-75 years were included. Hemiplegic patients with shoulder pain formed the first group, while those without shoulder pain formed the second group. Shoulder pain was assessed using the Visual Analog Scale (VAS), shoulder range of motion with the Senso4Motion device, and balance level with both the Berg Balance Scale and Senso4Motion.

DETAILED DESCRIPTION:
Hemiplegia is one of the most frequent clinical outcomes after stroke and is commonly accompanied by shoulder problems, which are a major cause of impaired biomechanics. Shoulder function plays a key role in transfers, maintaining postural stability during ambulation, and ensuring effective hand and self-care functions. Impaired shoulder biomechanics may cause a feeling of insecurity, abnormal gait disturbances, and balance deficits.

The primary objective of this study is to evaluate the effect of shoulder problems on balance in hemiplegic patients. Inclusion criteria were: first-ever diagnosis of stroke, Mini Mental State Examination score ≥24, voluntary participation, literacy, absence of visual impairment, and age between 40-75 years. Participants signed informed consent forms and completed a demographic data form including sex, age, height, weight, education level, medical and family history, smoking status, other comorbidities, affected side, and duration of hemiplegia.

Hemiplegic patients were divided into two groups: those with shoulder pain and those without. Shoulder pain was assessed using the Visual Analog Scale (VAS). Shoulder joint range of motion was measured with the Senso4Motion device. Balance performance was evaluated using the Berg Balance Scale and the Senso4Motion system. By comparing patients with and without shoulder pain, this study aims to clarify the impact of shoulder problems on post-stroke balance, thereby contributing to rehabilitation strategies and improving functional outcomes

ELIGIBILITY:
Inclusion Criteria:

Voluntary participation with signed informed consent Ability to read and write Age between 40 and 80 years First-ever stroke diagnosis Stable vital signs

Exclusion Criteria:

Diagnosis of any neurological or psychiatric disorder other than stroke Presence of visual or speech impairments History of more than one stroke

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of hemiplegic patients aged 40 to 80 years who experienced a first-ever stroke. Participants were recruited from [insert hospital/clinic name, e.g., Istanbul Aydın University affiliated hospitals/outpatient clinics]. Eligible patients had stable vital signs, adequate cognitive function (MMSE ≥ 24), and the ability to read and write. Patients were divided into subgroups according to the presence or absence of shoulder problems
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-07 (Estimated); Primary Completion 2025-10-07 (Estimated); Study Completion 2025-11-07 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain (Visual Analog Scale - VAS) | At baseline (single assessment)
  Shoulder pain will be assessed using a 10-cm Visual Analog Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst imaginable pain".

SECONDARY OUTCOMES:
Berg Balance Scale | at baseline (single assesment)
  Balance performance will be evaluated using the Berg Balance Scale (BBS). Scores range from 0 to 56, with higher scores indicating better balance ability.
Eularia Health - Eularia Lab | at baseline (single assesment)
  Balance performance will also be assessed using the Eularia Health - Euralia Lab system, which provides objective measurements of postural stability, movement parameters, and dynamic balance control.

CONTACTS AND LOCATIONS:
Overall Officials: GÖKHAN ÖZKOÇAK, M.D., Study Chair — İSTANBUL AYDIN UNIVERSITY; İBRAHİM HALİL URAL, M.D, Study Chair — İstanbul Beykent Unıversıty; ARZU DİNÇ YAVAŞ, M.D, Study Chair — Istanbul Aydın University; eda salgut, PT, Principal Investigator — İSTANBUL AYDIN UNIVERSITY
Locations (1):
- İstanbul Aydın Unıversity, Istanbul, KÜÇÜKÇEKMECE, Turkey (Türkiye)